CLINICAL TRIAL: NCT01959542
Title: Early Changes in Multiparametric MRI in Response to Neoadjuvant Androgen Deprivation and External Beam Radiation Therapy for Prostate Cancer
Brief Title: Early Changes In Multiparametric MRI In Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fiona Fennessy, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-343; U01CA151261 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRIs and PSA Blood Test (Experimental): * Visit 1 (8 weeks after starting ADT): PSA blood test and prostate MRI
  * Visit 2 (6 weeks after starting EBRT): PSA blood test and prostate MRI
  * Visit 3 (on last day of EBRT): PSA blood test
  * Visit 4 (6 months after starting ADT): PSA blood test and prostate MRI
  Interventions: Device: MRI; Other: PSA Blood Test

INTERVENTIONS:
Device: MRI
Other: PSA Blood Test — Serum PSA will also be subsequently checked on the same day as each follow-up MR is performed, i.e. TP 1, 2 and 3, and right after finishing EBRT. 1-2 mls of blood will be sampled per blood test.

SUMMARY:
In this research study, the investigators are trying to determine if there are measurable changes in prostate MRI that will help predict those who will or will not respond to Androgen Deprivation Therapy (ADT) and External Beam Radiation Therapy (EBRT) The first baseline prostate MRI prior to the start of treatment is standard of care. The participant's ADT/EBRT treatment is also standard of care, as advised by their doctor. It is the 3 follow up prostate MRIs during ADT/EBRT treatment, and 4 follow up serum PSA levels that are part of this research study.

DETAILED DESCRIPTION:
If the participant chooses to take part in this research study, the participant will have 3 follow up prostate MRIs during a 6 month time period, while the participant is having their ADT/EBRT treatment. These follow-up prostate MRIs will use a standard imaging protocol without the use of an endorectal coil. The participant will also have a total of 4 blood samples to measure serum PSA. 1-2 mls (just less than ½ teaspoon) will be taken for each sample.

Research Study Plan

* Baseline Visit (routine standard of care screening visit): PSA blood test and prostate MRI
* Visit 1 (8 weeks after starting ADT): PSA blood test and prostate MRI
* Visit 2 (6 weeks after starting EBRT): PSA blood test and prostate MRI
* Visit 3 (on last day of EBRT): PSA blood test
* Visit 4 (6 months after starting ADT): PSA blood test and prostate MRI

Planned Follow-up: The investigator would like to keep track of the participant's prostate cancer status while they continue to see their doctor at DFCI. The investigators would like to do this by collecting the following data from the participant's medical records, to look at long-term outcome of their ADT/EBRT treatment.

* PSA values
* Clinical results of your treatment. The investigator will not contact the participant to obtain this information.

ELIGIBILITY:
Inclusion Criteria:

* Adult males with unfavorable intermediate- to high-risk localized disease, defined as having one of the following three categories, Clinical or radiographic T2b-T4 primary tumor or Gleason score 7-10 in any core, or PSA ≥ 10 prior to initiation of therapy
* Patients are deemed suitable for therapy with ADT and EBRT.
* Subjects must to able to provide informed written consent prior to study entry.

Exclusion Criteria:

* The standard exclusion criteria for MRI exams will apply which include patients with pacemakers, non-compatible intra-cranial vascular clips, inner ear implants, and severe claustrophobia.
* Patients who because of age, general medical or psychiatric condition, or physiologic status unrelated to the presence of prostate cancer are unlikely to be candidates for repeat MRIs, or cannot give valid informed consent.
* Patients unwilling or unable to undergo the multiparametric MRI exam (non-endorectal coil).
* Patients with a history of allergic reaction to latex or Gadolinium containing intravenous contrast agents.
* Individuals with renal disease or other contraindications to gadolinium will be excluded. The BWH standard MRI contrast screening criteria will be used to establish renal status.
* Patients who have had prior prostatectomy or prior androgen therapy.
* Patients with hip implant or any other metallic implant or device that results in significant distortion of the local magnetic field and compromise of the quality of the multiparametric MRI data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Fennessy, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: All enrolled patients undergo PSA sampling and prostate MRI. No control arm.
Period: Overall Study
Arm/Group | Single Arm
Started (3 patients withdrew after initial consent.) | 15
Evaluable at Visit 1 | 12
Evaluable at Visit 2 | 12
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- MRIs and PSA Blood Test: * Visit 1 (8 weeks after starting ADT): PSA blood test and prostate MRI
  * Visit 2 (6 weeks after starting EBRT): PSA blood test and prostate MRI
  * Visit 3 (on last day of EBRT): PSA blood test
  * Visit 4 (6 months after starting ADT): PSA blood test and prostate MRI
  MRI
  PSA Blood Test: Serum PSA will also be subsequently checked on the same day as each follow-up MR is performed, i.e. TP 1, 2 and 3, and right after finishing EBRT. 1-2 mls of blood will be sampled per blood test.
  Androgen Deprivation Therapy (ADT): Patients will receive ADT as part of their standard clinical care, as determined by their clinician.
  External Beam Radiation Therapy (EBRT): Patients will receive EBRT as part of their standard clinical care, as determined by their clinician.
Arm/Group | MRIs and PSA Blood Test
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: mean] | 70.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
baseline PSA [Mean (Standard Deviation); unit: ng/ml] | 24.75 (32.01)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between MRI Parameter at Visit 1 and Nadir PSA
Description: Pearson correlation coefficient between MRI parameters at visit 1 and nadir PSA
Time Frame: 2 months after starting ADT (Visit 1)
Population: 12 patients enrolled. For one patient, data was not extracted from the MRI due to artifact.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Single Arm
Number analyzed (Participants) | 11
correlation coefficient | -0.53 [-0.86 to 0.10]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other — Pearson's product-moment correlation; p = 0.09, Pearson's product-moment correlation; Pearson's product-moment correlation = -0.53, 95% CI 2-sided [-086 to 0.10]

2. Secondary Outcome: Correlation Between MRI Parameter at Visit 2 With Nadir PSA
Description: Pearson correlation coefficient between MRI parameters at visit 2 with nadir PSA
Time Frame: 6 weeks after starting EBRT (Visit 2)
Measure: Number (95% Confidence Interval); unit: Pearson correlation coefficient
Groups:
- MRIs and PSA Blood Test: All enrolled patients undergo PSA sampling and prostate MRI. No control arm.
Arm/Group | MRIs and PSA Blood Test
Number analyzed (Participants) | 12
Pearson correlation coefficient | -0.62 [-0.88 to -0.08]
Statistical Analysis 1: Comparison: MRIs and PSA Blood Test; Test type: Other; p = 0.03, Pearson's product-moment correlation; Pearson's product moment correlation; Pearson's product-moment correlation = -0.62, 95% CI 2-sided [-0.62 to -0.15]

ADVERSE EVENTS:
Time Frame: During and immediately after the MRIs.
Description: Adverse events included any serious events related to the MRI exam. Expected adverse events from MRI are not serious and include claustrophobia while in the MRI magnet, a warming sensation while in the MRI magnet, or infiltration of intravenous contrast in the subcutaneous tissues at the time of its administration.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT01959542/Prot_SAP_000.pdf